CLINICAL TRIAL: NCT04246086
Title: A Phase Ib/II, Open-Label, Multicenter Study With a Non-Randomized Stage Evaluating the Safety, Pharmacokinetics, and Efficacy of Mosunetuzumab Plus Lenalidomide (+Len), and a Randomized Stage Evaluating the Safety, Tolerability, and Pharmacokinetics of SC Versus IV Mosunetuzumab + Len in Patients With Follicular Lymphoma
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, and Efficacy of Mosunetuzumab + Lenalidomide (+Len), and the Safety, Tolerability, and Pharmacokinetics of SC Versus IV Mosunetuzumab + Len in Participants With Follicular Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CO41942; 2019-004291-20 (EudraCT Number)
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — tocilizumab; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Intravenous (IV) Mosunetuzumab + Lenalidomide (Non-randomized) (Experimental): Participants will receive treatment with IV mosunetuzumab plus lenalidomide for 12 cycles total (cycle length = 21 days for Cycle 1, 28 days from Cycle 2 onward)
  Interventions: Drug: Mosunetuzumab (IV); Drug: Tocilizumab; Drug: Lenalidomide
- Subcutaneous (SC) Mosunetuzumab + Lenalidomide (Non-randomized) (Experimental): Participants will receive treatment with SC mosunetuzumab plus lenalidomide for 12 cycles total (cycle length = 21 days for Cycle 1, 28 days from Cycle 2 onward). Participants that have received complete metabolic response (CMR) or partial metabolic response (PMR) after 12 cycles of induction therapy with mosunetuzumab + lenalidomide will receive maintenance therapy with SC mosunetuzumab every 8 weeks (Q8W) for an additional 9 cycles.
  Interventions: Drug: Tocilizumab; Drug: Lenalidomide
- Arm A: IV Mosunetuzumab + Len (Randomized) (Experimental): Participants will receive treatment with IV mosunetuzumab plus lenalidomide for 12 cycles total (cycle length = 21 days for Cycle 1, 28 days from Cycle 2 onward)
  Interventions: Drug: Mosunetuzumab (IV); Drug: Lenalidomide
- Arm B: SC Mosunetuzumab + Len (Randomized) (Experimental): Participants will receive treatment with SC mosunetuzumab plus lenalidomide for 12 cycles total (cycle length = 21 days for Cycle 1, 28 days from Cycle 2 onward)
  Interventions: Drug: Lenalidomide; Drug: Mosunetuzumab (SC)

INTERVENTIONS:
Drug: Mosunetuzumab (IV) — Participants will receive IV mosunetuzumab as defined by the study protocol
  Other Names: RO7030816
  Arms: Arm A: IV Mosunetuzumab + Len (Randomized); Intravenous (IV) Mosunetuzumab + Lenalidomide (Non-randomized)
Drug: Tocilizumab — Participants will receive IV tocilizumab as needed for adverse reactions as defined by the study protocol
  Other Names: RO4877533
  Arms: Intravenous (IV) Mosunetuzumab + Lenalidomide (Non-randomized); Subcutaneous (SC) Mosunetuzumab + Lenalidomide (Non-randomized)
Drug: Lenalidomide — Participants will receive oral lenalidomide as defined by the study protocol
Drug: Mosunetuzumab (SC) — Participants will receive SC mosunetuzumab as defined by the study protocol
  Other Names: RO7030816
  Arms: Arm B: SC Mosunetuzumab + Len (Randomized)

SUMMARY:
This study will evaluate the safety, efficacy, pharmacokinetics, and immunogenicity of mosunetuzumab (Mosun) + lenalidomide (Len) (Mosun + Len) in participants with follicular lymphoma (FL). This study will also compare the pharmacokinetics, pharmacodynamics, safety, efficacy, and immunogenicity of IV mosunetuzumab + len vs subcutaneous (SC) mosunetuzumab + len.

ELIGIBILITY:
Inclusion Criteria

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* R/R FL after treatment with at least one prior systemic lymphoma therapy, which includes prior immunotherapy or chemoimmunotherapy
* Previously untreated participants with FL must require systemic therapy assessed by investigator based on the Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria and have a Follicular Lymphoma International Prognostic Index (FLIPI) score of 2-5
* Histologically documented FL of Grade 1, 2, or 3a, and that expresses CD20 at time of diagnosis as determined by the local laboratory
* Fluorodeoxyglucose avid lymphoma (i.e., positron emission tomography (PET) positive lymphoma)
* At least one bi dimensionally measurable nodal lesion (>1.5 cm in its largest dimension by PET- computed tomography (CT) scan), or at least one bi dimensionally measurable extranodal lesion (>1.0 cm in its largest dimension by PET-CT scan)
* Availability of a representative tumor specimen and the corresponding pathology report for confirmation of the diagnosis of FL
* Adequate hematologic function (unless due to underlying lymphoma, per the investigator) as defined by the protocol
* Negative HIV test at screening, with the following exception: Individuals with a positive HIV test at screening are eligible provided they are stable on antiretroviral therapy for at least 4 weeks, have a CD4 count ≥ 200/mL, have an undetectable viral load, and have not had a history of opportunistic infection attributable to AIDS within the last 12 months
* Normal laboratory values (unless due to underlying lymphoma) as defined by the protocol
* Agreement to comply with all local requirements of the Len risk minimization plan
* For women of childbearing potential: agreement to remain abstinent or use two adequate methods of contraception, including at least one method with a failure rate of < 1% per year, for at least 28 days prior to Day 1 of Cycle 1, during the treatment period, and for at least 12 months after the final dose of glofitamab, 28 days after the last dose of Len, 18 months after the last dose of G, 3 months after the final dose of tocilizumab, and 3 months after the final dose of Mosun. Women must refrain from donating eggs during this same period
* For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm, with female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 2 months after the final dose of glofitamab, 28 days after last dose of Len, 18 months after the last dose of G, 3 months after the final dose of tocilizumab, and 3 months after the final dose of Mosun

Exclusion Criteria

* Any history of Grade 3b FL
* Suspicion or clinical evidence of transformed lymphoma at enrollment by investigator assessment
* Any history of disease transformation and/or diffuse large B-cell lymphoma (DLBCL)
* Documented refractoriness to an obinutuzumab monotherapy containing regimen in glofitamab-containing treatment combination
* Active or history of central nervous system (CNS) lymphoma or leptomeningeal infiltration
* Documented refractoriness to lenalidomide, defined as no response (partial response (PR) or complete response (CR)) within 6 months of therapy
* Prior standard or investigational anti-cancer therapy as specified by the protocol
* Clinically significant toxicity (other than alopecia) from prior treatment that has not resolved to Grade <=2 prior to Day 1 of Cycle 1
* Known history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterans), drug-induced pneumonitis or evidence of active pneumonitis on screening chest CT scan
* Treatment with systemic immunosuppressive medications, including, but not limited to, prednisone, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents within 2 weeks prior to Day 1 of Cycle 1
* History of solid organ transplantation
* History of severe allergic or anaphylactic reaction to humanized, chimeric or murine MAbs
* Known sensitivity or allergy to murine products
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the glofitamab, Mosun, G, Len, or thalidomide formulation, including mannitol
* History of erythema multiforme, Grade >=3 rash, or blistering following prior treatment with immunomodulatory derivatives
* Known history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis or evidence of active pneumonitis on screening chest CT scan
* Known active bacterial, viral, fungal, or other infection, or any major episode of infection requiring treatment with IV antibiotics within 4 weeks of Day 1 of Cycle 1
* Known or suspected chronic active Epstein-Barr virus infection or hemophagocytic syndrome
* Known history of macrophage activating syndrome (MAS) or hemophagocytic lymphohistiocytosis (HLH)
* Active Hepatitis B and Hepatitis C infection or autoimmune disease requiring treatment
* Prior allogenic hematopoietic stem cell transplant
* Known history of HIV positive status
* History of progressive multifocal leukoencephalopathy
* Administration of a live, attenuated vaccine within 4 weeks before first dose of study treatment or anticipation that such a live attenuated vaccine will be required during the study
* Other malignancy that could affect compliance with the protocol or interpretation of results
* Prior allogenic hematopoietic stem cell transplant (HSCT)
* Contraindication to treatment for thromboembolism prophylaxis
* Grade >=2 neuropathy
* Evidence of any significant, uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including, but not limited to significant cardiovascular disease or significant pulmonary disease
* Major surgical procedure other than for diagnosis within 28 days prior to Day 1 of Cycle 1 Day 1 or anticipation of a major surgical procedure during the course of the study
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Inadequate hematologic function
* Any of the following abnormal laboratory values
* Pregnant or lactating or intending to become pregnant during the study
* Life expectancy < 3 months
* Unable to comply with the study protocol, in the investigator's judgment
* History of illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's or Medical Monitor's judgment, precludes the patient's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2030-10-15 (Estimated); Study Completion 2030-10-15 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities (DLTs) | Cycle 2 Days 1-28 (cycle length = 28 days)
Percentage of Participants with Adverse Events | From baseline to 90 days after the last dose of study drug
Cumulative Area under the Curve over Cycles 1-3 (AUC1-3) of Mosunetuzumab | Day 1 - Day 78
Serum Trough Concentration at Steady State Approximated by Cycle 4 (Ctrough, c4) of Mosunetuzumab | Day 106
Overall Response Rate (ORR) as Determined by the Independent Review Committee (IRC) | Up to the end of Cycle 12 (cycle length = 28 days)

SECONDARY OUTCOMES:
Complete Response Rate (CRR) as determined by the investigator (non-randomized stage) | Up to the end of Cycle 12 (cycle length = 28 days)
CRR as determined by Independent Review Committee (IRC) (randomized stage) | Up to the end of Cycle 12 (cycle length = 28 days)
Objective Response Rate (ORR) as determined by the investigator (non-randomized stage) | Up to the end of Cycle 12 (cycle length = 28 days)
ORR as determined by IRC (randomized stage) | Up to the end of Cycle 12 (cycle length = 28 days)
Duration of Response (DOR) as determined by the investigator (non-randomized stage) | From the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, up to the end of Cycle 8 (cycle length = 28 days)
DOR as determined by IRC (randomized stage) | From the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, up to the end of Cycle 8 (cycle length = 28 days)
Duration of Complete Reponse (DOCR) as determined by the investigator (non-randomized stage) | From the first occurrence of a documented complete response (CR) to disease progression, relapse, or death from any cause, whichever occurs first, up to the end of Cycle 12 (cycle length = 28 days)
DOCR as determined by IRC (randomized stage) | From the first occurrence of a documented complete response (CR) to disease progression, relapse, or death from any cause, whichever occurs first, up to the end of Cycle 12 (cycle length = 28 days)
Percentage of Participants with AEs (Arms A and B) | From baseline to 90 days after the last dose of study drug
Minimum Serum Concentration (Cmin) of Mosunetuzumab | At pre-defined intervals from Cycle 1 Day 1 through follow up (2 years after last treatment)
Maximum Serum Concentration (Cmax) of Mosunetuzumab | At pre-defined intervals from Cycle 1 Day 1 through follow up (2 years after last treatment)
Cumulative AUC Over Cycles 1-2 (AUCc1-2) of Mosunetuzumab (Arms A and B) | Day 1 - Day 50
Serum Trough Concentration in Cycle 2 (Ctrough, c2) of Mosunetuzumab (Arms A and B) | Day 50
AUC at Steady State (AUCss) (Arms A and B) | Cycle 4 (cycle length = 28 days)
Percentage of Participants with ADAs to Mosunetuzumab | At pre-defined intervals from baseline through follow-up (2 years after last treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- United States (12):
  - City of Hope National Medical Center, Duarte, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Mary Bird Perkins Cancer Ctr, Baton Rouge, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Hillcrest Hospital, Mayfield Heights, Ohio
  - Rhode Island Hematology/Oncology Program, Woonsocket, Rhode Island
  - Tennessee Oncology;Chattanooga Oncology & Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology PLLC - Franklin, Franklin, Tennessee
  - Swedish Medical Center, Seattle, Washington
- China (6):
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjing
  - The First Affiliated Hospital of Xiamen University, Xiamen
- France (6):
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - CHU Montpellier, Montpellier
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - Institut Claudius Regaud, Toulouse
- Spain (4):
  - Hospital Universitario Vall d Hebron, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz., Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Complejo Asistencial Universitario de Salamanca, Salamanca
- United Kingdom (5):
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing